CLINICAL TRIAL: NCT02665429
Title: A Quality Improvement Project to Investigate Individual Provider Variation in Opioid Prescribing From the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: UMass Memorial Health (Other)
Responsible Party: Principal Investigator, Sean Michael, Emergency Medicine Administrative Leadership Fellow, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H00009241
Record Dates: First submitted 2016-01-20; First posted 2016-01-27 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Analgesics, Opioid; Delivery of Health Care; Drug Prescribing; Over Prescribing; Prescribing Patterns, Physician; Practice Management, Medical; Practice Guidelines as Topic
Keywords: Emergency Medicine
MeSH Terms: interventions — Diagnostic Self Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Providers who are subject only to the routine implementation of clinical practice guidelines without additional experimental intervention
- Intervention (Experimental): Providers who are subject to routine clinical practice guideline implementation AND receive provider's own individual prescribing data profile intervention ("Individual prescribing data profile and self-assessment")
  Interventions: Behavioral: Individual prescribing data profile and self-assessment

INTERVENTIONS:
Behavioral: Individual prescribing data profile and self-assessment — Prior to receiving his or her individual data profile, each provider in the intervention group will be asked to identify his or her self-assessment of his or her own opioid prescribing practices. Immediately after providing self-perception data, providers will be provided with their true profile data with a visual display of where they fall within the distribution of their peers. All peer data are de-identified.
  Arms: Intervention

SUMMARY:
This is a study of emergency physicians' prescribing patterns related to opioid (narcotic) medications. We are trying to determine whether giving providers access to their own prescribing data influences their prescribing patterns.

DETAILED DESCRIPTION:
Opioid misuse is a known public safety threat and public health problem, both nationwide and in the Commonwealth of Massachusetts. As a part of these efforts, Emergency Department (ED) outpatient prescriptions have been identified as a potential area for improvement. The Massachusetts Hospital Association (MHA), in conjunction with other stakeholders, developed a set of recommendations to address opioid management and prescribing within the ED setting.

This study is timed to coincide with the rollout by UMassMemorial Health Care of a system-wide opioid prescribing practice guideline/policy which mirrors the Massachusetts Hospital Association's guideline. This rollout provides a unique opportunity for a natural experiment related to provider prescribing practices.

This is a quality improvement project with two primary objectives:

* Improve understanding of physician practice patterns related to emergency department (ED) opioid prescribing
* Evaluate the effectiveness of providing individual clinician profile data in influencing behavior change among ED providers, as it relates to their opioid prescribing patterns

There are two corresponding specific aims:

* Quantitatively describe the current state of opioid prescribing by ED clinicians at four UMass Memorial EDs (using prescriptions generated within the ED electronic health information system between February 2014 and the study implementation date). Descriptive statistics being considered for feasibility of study include:
* Number of opioid prescriptions per hundred patients seen
* Percentage of total prescriptions written that are opioids
* Mean or median quantity of pills dispensed per opioid prescription
* Number of prescriptions for long-acting opioid formulations
* Evaluate the effect on prescribing practices of providing individual clinicians with their profile data to illustrate their personal opioid prescribing patterns, relative to the de-identified distribution for all other clinicians in the ED group

This project is timed to coincide with the separately planned implementation of a system-wide opioid prescribing guideline. The guideline implementation is an independent event, but we feel that it presents a unique opportunity for a simultaneous experimental intervention to assess whether providing clinicians with their individual data alters their prescribing practices beyond any effect achieved simply by being subject to the new guideline. Data collected from the electronic medical record and clinician self-reported data about their perceptions of their prescribing practices will be used to evaluate both the effect of the guideline implementation (i.e. comparison of prescribing patterns for all clinicians before and after guideline implementation) and the combined effect of guideline implementation plus individual profile intervention (i.e. comparisons across intervention versus control groups).

ELIGIBILITY:
Inclusion Criteria:

* Provider who practices Emergency Medicine in one or more of four UMass-affiliated EDs (UMassMemorial Medical Center, Marlborough Hospital, and Clinton Hospital), including attending physicians, resident physicians, and advanced practice providers (PAs and NPs).
* Have placed at least one electronic prescription for a medication of interest (namely opioids) in the PulseCheck electronic medical record system during the 12 months prior to the implementation of the opioid guidelines
* Be actively practicing in a UMass-affiliated ED at time of implementation of the guidelines

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Change in number of opioid prescriptions per hundred patients seen | Pre-intervention baseline compared to 1, 2, 3, 6, 9, 12 months post-intervention

SECONDARY OUTCOMES:
Change in percentage of total prescriptions written that are opioids | Pre-intervention baseline compared to 1, 2, 3, 6, 9, 12 months post-intervention
Change in median quantity of pills dispensed per opioid prescription | Pre-intervention baseline compared to 1, 2, 3, 6, 9, 12 months post-intervention
Change in number of prescriptions for long-acting opioid formulations | Pre-intervention baseline compared to 1, 2, 3, 6, 9, 12 months post-intervention

OTHER OUTCOMES:
Self-assessment of decile for number of opioid prescriptions per hundred patients seen | Once, at time of enrollment
  The provider's self-assessment of their decile of number of opioid prescriptions per hundred patients seen, compared to their peers
Self-assessment of decile for percentage of total prescriptions written that are opioids | Once, at time of enrollment
  The provider's self-assessment of their decile of their percentage of total prescriptions written that are opioids, compared to their peers
Self-assessment of decile for median quantity of pills dispensed per opioid prescription | Once, at time of enrollment
  The provider's self-assessment of their decile of their median quantity of pills dispensed per opioid prescription, compared to their peers
Self-assessment of decile for number of prescriptions for long-acting opioid formulations | Once, at time of enrollment
  The provider's self-assessment of their decile of their number of prescriptions for long-acting opioid formulations, compared to their peers

CONTACTS AND LOCATIONS:
Overall Officials: Sean Michael, MD, Principal Investigator — UMass Memorial Health
Locations (3):
- United States (3):
  - UMass Clinton Hospital, Clinton, Massachusetts
  - UMass Memorial Marlborough Hospital, Marlborough, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No